CLINICAL TRIAL: NCT00414050
Title: A Study to Assess the Safety, Tolerability, and Immunogenicity of 2 Antigen Doses of Recombinant Hepatitis B Vaccine Manufactured With a Modified Process Administered to Healthy Infants at 2, 4, and 6 Months of Age
Brief Title: A Study of 2 Doses of a Hepatitis B Vaccine (V232 RECOMBIVAX HB) in Healthy Infants (V232-057)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V232-057; 2006_053; 2006-001638-42 (EudraCT Number)
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Results first posted 2009-04-14 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines; Recombivax HB; Engerix-B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Modified Process Hepatitis B vaccine 5 μg (Experimental): Infants received a primary series of 3 doses of experimental vaccine (5 μg per dose) at 2, 4 and 6 months of age.
  Interventions: Biological: Modified Process Hepatitis B Vaccine (Experimental)
- RECOMBIVAX HB™ Hepatitis B Vaccine (Active Comparator): Infants received a primary series of 3 doses of currently licensed vaccine (5 μg per dose) at 2, 4 and 6 months of age.
  Interventions: Biological: Hepatitis B Vaccine (Recombinant)
- Modified Process Hepatitis B vaccine 10 μg (Experimental): Infants received a primary series of 3 doses of experimental vaccine (10 μg per dose) at 2, 4 and 6 months of age.
  Interventions: Biological: Modified Process Hepatitis B Vaccine (Experimental)
- ENGERIX-B® (Active Comparator): Infants received a primary series of 3 doses of currently licensed vaccine (10 μg per dose) at 2, 4 and 6 months of age.
  Interventions: Biological: Hepatitis B Vaccine (Recombinant)

INTERVENTIONS:
Biological: Modified Process Hepatitis B Vaccine (Experimental) — Modified Process Hepatitis B Vaccine given intramuscularly (IM) in 3 injections of 5 ug (micrograms)/0.5 mL each over 4 months (Modified Process Hepatitis B vaccine 5 μg arm). Modified Process Hepatitis B Vaccine given IM in 3 Injections of 10 ug (micrograms)/0.5 mL each over 4 months (Modified Process Hepatitis B vaccine 10 μg arm).
  Arms: Modified Process Hepatitis B vaccine 10 μg; Modified Process Hepatitis B vaccine 5 μg
Biological: Hepatitis B Vaccine (Recombinant) — RECOMBIVAX HB™ (currently licensed product) given IM in 3 Injections of 5 ug/0.5 mL each over 4 months.
  Other Names: RECOMBIVAX HB™
  Arms: RECOMBIVAX HB™ Hepatitis B Vaccine
Biological: Hepatitis B Vaccine (Recombinant) — ENGERIX-B® (currently licensed product) given IM in 3 Injections of 10 ug/0.5 mL each over 4 months
  Other Names: ENGERIX-B®
  Arms: ENGERIX-B®

SUMMARY:
This study was conducted in healthy infants and will provide new immunogenicity and safety data for the modified process hepatitis B vaccine. This study was conducted to address the following: to evaluate the immunogenicity and safety data of the 5 microgram dose of the modified process hepatitis B vaccine compared with a 10 microgram dose of the modified process hepatitis B vaccine, to evaluate another dosing schedule of 2, 4, and 6 months, and to provide descriptive immunogenicity data of another marketed vaccine (ENGERIX-B®).

ELIGIBILITY:
Inclusion Criteria:

* Participant is a healthy infant approximately 2 months of age

Exclusion Criteria:

* Birth mother is a known carrier of hepatitis B virus or another known carrier has lived in close contact with the participant
* Participant's birth mother did not receive any prenatal care
* Participant has previous history of hepatitis B infection
* Participant has been vaccinated against hepatitis B or birth mother was vaccinated within 6 months before birth of participant
* Participant has had a fever within 72 hours of study start
* Participant has received any blood-derived product or birth mother received blood-derived product within 6 months of birth of participant

Ages: 2 Months to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1718 (Actual)
Dates: Start 2006-10-06 (Actual); Primary Completion 2007-10-22 (Actual); Study Completion 2007-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Vesikari T, Martin JC, Liss CL, Liska V, Schodel FP, Bhuyan PK. Safety and immunogenicity of a modified process hepatitis B vaccine in healthy infants. Pediatr Infect Dis J. 2011 Jul;30(7):e109-13. doi: 10.1097/INF.0b013e31821ed1a4. PMID 21552183

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15-Nov-2006 (First Participant Enrolled in Study) to 24-Oct-2007 (Last Participant had their Last Visit). Last participant completed follow-up: 16-Oct-2007.This study was conducted at 15 sites; 14 in Finland and 1 in Norway.
Groups:
- Modified Process Hepatitis B Vaccine 5 µg (Micrograms): Infants received a primary series of 3 doses of experimental vaccine (5 μg per dose) at 2, 4 and 6 months of age.
- RECOMBIVAX™ Hepatitis B Vaccine: Infants received a primary series of 3 doses of currently licensed vaccine (5 μg per dose) at 2, 4 and 6 months of age.
- Modified Process Hepatitis B Vaccine 10 µg: Infants received a primary series of 3 doses of experimental vaccine (10 μg per dose) at 2, 4 and 6 months of age.
Period: Overall Study
Arm/Group | Modified Process Hepatitis B Vaccine 5 µg (Micrograms) | RECOMBIVAX™ Hepatitis B Vaccine | Modified Process Hepatitis B Vaccine 10 µg | ENGERIX-B®
Started | 431 | 427 | 429 | 431
Received Vaccination 1 | 431 | 426 | 429 | 431
Received Vaccination 2 | 425 | 421 | 425 | 425
Received Vaccination 3 | 424 | 419 | 425 | 424
Completed | 422 | 419 | 423 | 423
Not Completed | 9 | 8 | 6 | 8
Not completed — Adverse Event | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 2 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 5 | 3 | 2 | 4
Not completed — Subject discontinued for other reason | 1 | 2 | 2 | 1
Not completed — Subject Moved | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Process Hepatitis B Vaccine 5 µg (Micrograms) | RECOMBIVAX™ Hepatitis B Vaccine | Modified Process Hepatitis B Vaccine 10 µg | ENGERIX-B® | Total
Number analyzed (Participants) | 431 | 427 | 429 | 431 | 1718
Age, Continuous [Mean (Standard Deviation); unit: days] | 63.2 (10.18) | 62.9 (10.15) | 63.3 (9.83) | 62.8 (9.81) | 63.1 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 217 | 208 | 201 | 816
  Male | 241 | 210 | 221 | 230 | 902

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Seroresponders to the Modified Process Hepatitis B Vaccine (5 μg and 10 μg Dose), RECOMBIVAX HB™ Hepatitis B Vaccine (Currently Licensed Vaccine), and ENGERIX-B®
Description: The percentage of participants as measured by Seroresponse. Seroresponse was defined as anti-hepatitis B surface antibodies greater than or equal to 10 milli-International Units (mIU)/mL. Success on the primary immunogenicity hypothesis required demonstrating an adequate anti-HBs seroprotection rate response for either modified process hepatitis B 5 μg vaccine or RECOMBIVAX HB™. Specifically, the lower bound of the multiplicity adjusted 95% confidence interval (CI) on the seroprotection rate for either vaccine was required to be above 90.0%.
Time Frame: 7 months of age (1 month after 3 doses)
Population: Participants who follow the protocol, do not have major protocol deviations and have post-vaccination serology within specified day ranges.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Modified Process Hepatitis B Vaccine 5 µg (Micrograms) | RECOMBIVAX™ Hepatitis B Vaccine | Modified Process Hepatitis B Vaccine 10 µg | ENGERIX-B®
Number analyzed (Participants) | 405 | 406 | 398 | 400
Percentage of participants | 99.3 [98.3 to 100] | 98.5 [97.2 to 99.8] | 100 [99.9 to 100] | 99.5 [98.7 to 100]

2. Secondary Outcome: Antibody to Hepatitis B Surface Antigen Geometric Mean Titer (Anti-HBs GMT) Responses for Modified Process Vaccine (5 μg and 10 μg), RECOMBIVAX™ Hepatitis B (Currently Licensed Vaccine), and ENGERIX-B®
Description: Geometric Mean Titer - Antibody titer is a laboratory test that measures the presence and amount of antibodies in blood.
Time Frame: 7 months of age (1 month after 3 doses)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Modified Process Hepatitis B Vaccine 5 µg (Micrograms) | RECOMBIVAX™ Hepatitis B Vaccine | Modified Process Hepatitis B Vaccine 10 µg | ENGERIX-B®
Number analyzed (Participants) | 405 | 406 | 398 | 400
mIU/mL | 748.2 [672.0 to 833.1] | 376.8 [331.4 to 428.5] | 981.5 [891.0 to 1081.2] | 556.6 [491.8 to 629.9]
Statistical Analysis 1: Comparison: Modified Process Hepatitis B Vaccine 5 µg (Micrograms) vs RECOMBIVAX™ Hepatitis B Vaccine; Comparison of Induced (effected) Geometric Mean Titer for the Modified Hepatitis B Process Vaccine and RECOMBIVAX Hepatitis B vaccine; Test type: Non-Inferiority or Equivalence — Modified Process Hepatitis B vaccine-5µg (micrograms) declared non-inferior to RECOMBIVAX HB™ if the lower bound of the 95% Confidence Interval for the ratio of Geometric Mean Titers (Modified Process Vaccine 5 micrograms/RECOMBIVAX HB™) was >= 0.67. The study had 98 percent power for this test, based on an assumption of true equality; Ratio of geometric means = 1.99, 95% CI 2-sided [1.69 to 2.35]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs): up to 5 months (entire study period); Systemic non-serious adverse events (NSAEs): up to 14 days after any vaccination; Injection-site NSAEs: up to 5 days after any vaccination
Description: All randomized participants with follow-up who received at least one dose of study vaccine. Below tables exclude one RECOMBIVAX HB participant who received 2 doses of RECOMBIVAX HB™ and 1 dose of modified process hepatitis B vaccine 10 μg, and one ENGERIX-B® participant who received 2 doses of ENGERIX-B® and 1 dose of RECOMBIVAX HB™.
Arm/Group | Modified Process Hepatitis B Vaccine 5 µg (Micrograms) | RECOMBIVAX™ Hepatitis B Vaccine | Modified Process Hepatitis B Vaccine 10 µg | ENGERIX-B®
Serious Adverse Events (participants affected / at risk) | 11/430 | 2/424 | 6/429 | 8/428
Other Adverse Events (participants affected / at risk) | 308/430 | 294/424 | 276/429 | 288/428
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified Process Hepatitis B Vaccine 5 µg (Micrograms) (N=430) | RECOMBIVAX™ Hepatitis B Vaccine (N=424) | Modified Process Hepatitis B Vaccine 10 µg (N=429) | ENGERIX-B® (N=428)
Nutritional condition abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden infant death syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Crying (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pyelonephritis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified Process Hepatitis B Vaccine 5 µg (Micrograms) (N=430) | RECOMBIVAX™ Hepatitis B Vaccine (N=424) | Modified Process Hepatitis B Vaccine 10 µg (N=429) | ENGERIX-B® (N=428)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (21) | 15 (18) | 17 (19) | 25 (26)
Conjunctivitis (Eye disorders) | 9 (11) | 14 (14) | 10 (10) | 22 (23)
Irritability (General disorders) | 114 (169) | 109 (157) | 91 (138) | 107 (139)
Pyrexia (General disorders) | 62 (78) | 57 (65) | 56 (68) | 53 (65)
Injection-site erythema (General disorders) | 128 (169) | 117 (160) | 116 (153) | 94 (124)
Injection-site pain (General disorders) | 79 (117) | 73 (96) | 60 (90) | 66 (92)
Injection-site induration (General disorders) | 25 (29) | 15 (19) | 24 (26) | 8 (9)
Injection-site swelling (General disorders) | 78 (109) | 85 (111) | 87 (110) | 65 (98)
Crying (Psychiatric disorders) | 41 (51) | 39 (49) | 39 (48) | 41 (48)
Diarrhoea (Gastrointestinal disorders) | 30 (37) | 26 (36) | 26 (31) | 18 (26)
Upper respiratory tract infection (Infections and infestations) | 32 (35) | 26 (27) | 25 (25) | 23 (25)
Rhinitis (Infections and infestations) | 53 (57) | 47 (54) | 59 (68) | 51 (57)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.